CLINICAL TRIAL: NCT01076530
Title: A Phase I Study of SAHA and Temozolomide in Children With Relapsed or Refractory Primary Brain or Spinal Cord Tumors
Brief Title: Vorinostat and Temozolomide in Treating Young Patients With Relapsed or Refractory Primary Brain Tumors or Spinal Cord Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02011; ADVL0819; CDR0000664388; COG-ADVL0819; U01CA097452 (NIH)
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Childhood Atypical Teratoid/Rhabdoid Tumor; Childhood Central Nervous System Choriocarcinoma; Childhood Central Nervous System Embryonal Tumor; Childhood Central Nervous System Germinoma; Childhood Central Nervous System Mixed Germ Cell Tumor; Childhood Central Nervous System Teratoma; Childhood Central Nervous System Yolk Sac Tumor; Childhood Choroid Plexus Tumor; Childhood Craniopharyngioma; Childhood Ependymoblastoma; Childhood Grade I Meningioma; Childhood Grade II Meningioma; Childhood Grade III Meningioma; Childhood High-grade Cerebellar Astrocytoma; Childhood High-grade Cerebral Astrocytoma; Childhood Infratentorial Ependymoma; Childhood Low-grade Cerebellar Astrocytoma; Childhood Low-grade Cerebral Astrocytoma; Childhood Medulloepithelioma; Childhood Mixed Glioma; Childhood Oligodendroglioma; Childhood Supratentorial Ependymoma; Extra-adrenal Paraganglioma; Recurrent Childhood Brain Stem Glioma; Recurrent Childhood Central Nervous System Embryonal Tumor; Recurrent Childhood Cerebellar Astrocytoma; Recurrent Childhood Cerebral Astrocytoma; Recurrent Childhood Ependymoma; Recurrent Childhood Medulloblastoma; Recurrent Childhood Pineoblastoma; Recurrent Childhood Spinal Cord Neoplasm; Recurrent Childhood Subependymal Giant Cell Astrocytoma; Recurrent Childhood Supratentorial Primitive Neuroectodermal Tumor; Recurrent Childhood Visual Pathway and Hypothalamic Glioma
MeSH Terms: conditions — Rhabdoid Tumor; Choroid Plexus Neoplasms; Astrocytoma; Oligodendroglioma; Paraganglioma, Extra-Adrenal; Familial ependymoma; Medulloblastoma; Spinal Cord Neoplasms; Optic Nerve Glioma | interventions — Vorinostat; Temozolomide

ARMS (1):
- Arm I (Experimental): Patients receive oral vorinostat and oral temozolomide once daily on days 1-5. Courses repeat every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vorinostat; Drug: temozolomide; Other: diagnostic laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: vorinostat
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Drug: temozolomide
  Other Names: SCH 52365; Temodal; Temodar; TMZ
Other: diagnostic laboratory biomarker analysis
Other: pharmacological study
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of vorinostat when given together with temozolomide in treating young patients with relapsed or refractory primary brain tumors or spinal cord tumors. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vorinostat may help temozolomide work better by making tumor cells more sensitive to the drug.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose and/or recommended phase II dose of vorinostat in combination with temozolomide in pediatric patients with relapsed or refractory primary CNS tumors.

II. To define and describe the toxicities of this regimen in these patients.

SECONDARY OBJECTIVES:

I. To preliminarily define the antitumor activity of this regimen within the confines of a phase I study.

II. To characterize the pharmacokinetic parameters of vorinostat in these patients.

III. To determine whether acetylated histones in peripheral blood mononuclear cells can be identified as a surrogate marker of the biologic effect of vorinostat at various treatment doses.

IV. To assess the feasibility of collecting and analyzing serum DNA for methylation of the MGMT promoter and describe the relationship between promoter methylation and clinical responses within the confines of this phase I study.

OUTLINE: This is a multicenter, dose-escalation study of vorinostat.

Patients receive oral vorinostat and oral temozolomide once daily on days 1-5. Courses repeat every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.

Patients may undergo blood sample collection periodically for pharmacokinetic and correlative laboratory studies by western blotting and MGMT promoter methylation assays.

After completion of study therapy, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CNS malignancy at original diagnosis or relapse

  * Histologic confirmation not required for patients with intrinsic brain stem tumors, optic pathway gliomas, or pineal tumors provided CSF or serum tumor markers, including alpha-fetoprotein orbeta-HCG, are elevated
  * Recurrent or refractory spinal cord tumors allowed
* Measurable or evaluable disease
* No known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Karnofsky performance status (PS) 50-100% (for patients > 16 years of age) OR Lansky PS 50-100% (for patients ≤ 16 years of age)

  * Neurological deficits must have been relatively stable for ≥ 1 week before study entry
  * Patients unable to walk due to paralysis, but who are up in a wheelchair, are considered ambulatory for the purpose of assessing performance status
* ANC ≥ 1,000/μL
* Platelet count ≥ 100,000/μL (transfusion independent, defined as no platelet transfusion within the past 7 days)
* Hemoglobin ≥ 8.0 g/dL (RBC transfusions allowed)
* Creatinine clearance or radioisotope GFR ≥ 70mL/min OR maximum serum creatinine based on age and/or gender as follows:

  * 0.6 mg/dL (1 year of age)
  * 0.8 mg/dL (2 to 5 years of age)
  * 1.0 mg/dL (6 to 9 years of age)
  * 1.2 mg/dL (10 to 12 years of age)
  * 1.5 mg/dL (males) or 1.4 mg/dL (females) (13 to 15 years of age)
  * 1.7 mg/dL (males) or 1.4 mg/dL (females) (≥ 16 years of age)
* Bilirubin ≤ 1.5 times upper limit of normal
* ALT ≤ 110 U/L
* Serum albumin ≥ 2 g/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to swallow capsules or liquid
* Seizure disorder allowed provided it is well controlled with nonenzyme-inducing anticonvulsants
* No pre-existing QTc ≥ 450 msec
* No uncontrolled infection
* No patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of study
* Fully recovered from prior chemotherapy, immunotherapy, or radiotherapy
* More than 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosourea)
* At least 7 days since prior hematopoietic growth factors
* At least 7 days since prior biologic agent (antineoplastic agent)
* At least 7 days or 3 half-lives, whichever is longer, since prior monoclonal antibodies
* More than 2 weeks since prior local palliative radiotherapy (small port)
* At least 6 months since prior total-body radiotherapy (TBI), craniospinal radiotherapy, or radiotherapy to ≥ 50% of the pelvis
* At least 6 weeks since other prior substantial bone marrow radiotherapy
* At least 3 months since prior stem cell transplantation or rescue (without TBI)

  * No evidence of active graft-vs-host disease
* At least 2 weeks since prior valproic acid
* No prior vorinostat
* Prior temozolomide allowed provided there was no progressive disease during or within 1 month after completion of treatment
* Concurrent corticosteroids allowed provided patient has been on a stable or decreasing dose for ≥ 7 days before study entry
* No other concurrent investigational drugs
* No other concurrent anticancer agents, including chemotherapy, radiotherapy, immunotherapy, or biologic therapy
* No concurrent enzyme-inducing anticonvulsants

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2010-02; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose defined as the maximum dose at which fewer than one-third of patients experience DLT using NCI CTCAE version 4.0 | 28 days
  In addition to determination of the MTD, a descriptive summary of all toxicities will be reported.
Pharmacokinetic parameters of vorinostat in combination with temozolomide | Pre-dose, 15 and 30 minutes, 1, 2, 4, 6, 8, and 24 hours
  The PK parameters will be summarized with simple summary statistics, including means, medians, ranges, and standard deviations (if numbers and distribution permit).

SECONDARY OUTCOMES:
Response assessed according to RECIST criteria | Up to 30 days
  Will be reported descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Trent Hummel, Principal Investigator — COG Phase I Consortium
Locations (9):
- United States (7):
  - Childrens Memorial Hospital, Chicago, Illinois
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Oregon Health and Science University, Portland, Oregon
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Canada (2):
  - Hospital for Sick Children, Toronto, Ontario
  - Hospital Sainte-Justine, Montreal, Quebec

REFERENCES:
- [Derived] Hummel TR, Wagner L, Ahern C, Fouladi M, Reid JM, McGovern RM, Ames MM, Gilbertson RJ, Horton T, Ingle AM, Weigel B, Blaney SM. A pediatric phase 1 trial of vorinostat and temozolomide in relapsed or refractory primary brain or spinal cord tumors: a Children's Oncology Group phase 1 consortium study. Pediatr Blood Cancer. 2013 Sep;60(9):1452-7. doi: 10.1002/pbc.24541. Epub 2013 Mar 28. PMID 23554030